CLINICAL TRIAL: NCT07119034
Title: Assessment of Oxidative Stress Parameters in Jordanian Pregnant Women With Preeclampsia
Brief Title: Assessment of Oxidative Stress Contents in Jordanian Pregnant Women With Preeclampsia
Acronym: Preeclampsia
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Collaborators: Al-Ahliyya Amman University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assistant professor of clinical Pharmacy, Al-Ahliyya Amman University
Other Study IDs: Al-Ahliyya Amman University; Preeclsmpsia (Registry Identifier: Al-Ahliyya Amman University); Preeclampsia (Other: Al-Ahliyya Amman University)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Preeclampsia (PE); Oxidative Stress
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples Without DNA — Blood samples were collected from the antecubital vein and processed at the TrueLab medical laboratory. The whole blood was initially collected in plain tubes, and subsequently centrifuged to obtain serum samples. Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) levels were measured. The remaining serum samples were stored at -80°C until analysis at AAU's clinical laboratory, utilizing Enzyme-linked immunosorbent assay (ELISA) for Thioredoxin and 4-Hydroxynonenal quantification, while malondialdehyde levels were measured using a colorimetric assay.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: control group comprising 45 healthy pregnant women
  Interventions: Diagnostic Test: Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)
- Preeclampsia group: Preeclampsia group 45 women with preeclampsia
  Interventions: Diagnostic Test: Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)

INTERVENTIONS:
Diagnostic Test: Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) — Blood samples were collected from the antecubital vein and processed at the TrueLab medical laboratory. The whole blood was initially collected in plain tubes, and subsequently centrifuged to obtain serum samples. Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) Thioredoxin and 4-Hydroxynonenal quantification, malondialdehyde levels

SUMMARY:
Preeclampsia, a widespread complication affecting pregnant women globally, necessitates a thorough investigation into the role of oxidative stress in its manifestation. This study aimed to assess the oxidative stress markers-malondialdehyde (MDA), 4-hydroxynonenal (4-HNE), and thioredoxin (Trx) in preeclamptic compared to healthy pregnant women

DETAILED DESCRIPTION:
Preeclampsia, a widespread complication affecting pregnant women globally, necessitates a thorough investigation into the role of oxidative stress in its manifestation. This study aimed to assess the oxidative stress markers-malondialdehyde (MDA), 4-hydroxynonenal (4-HNE), and thioredoxin (Trx) in preeclamptic compared to healthy pregnant women.

Methods: Ethical approval was obtained from Al-Ahliyya Amman University prior to starting the study. A total of 90 participants (45 preeclamptic pregnant women and 45 healthy pregnant women) were included in this study. Serum levels of total cholesterol (TC), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) were measured by HUMAN200 auto analyzer (Germany) using a homogeneous enzymatic colorimetric assay. A kit from GenoChem world was used to measure the MDA levels via a colorimetric analysis technique Sandwich enzyme-linked immunosorbent assay (ELISA) was used to determine the serum levels of Trx and 4-HNE.

Results: The results revealed significantly elevated levels of MDA and 4-HNE in preeclamptic women compared to their healthy counterparts (P<0.001). Although Trx levels did not differ significantly (P=0.29), marked distinctions were observed in LDL-C, TC, HDL-C, systolic and diastolic blood pressure (P<0.001). Preeclamptic women exhibited substantially higher LDL, TC, and blood pressure, and lower HDL.

Conclusion: This study highlights the correlation between elevated oxidative stress markers and an elevated risk of preeclampsia in pregnant women, which may suggest the impact of these markers in the pathogenesis of preeclampsia. These findings underscore the need for a nuanced understanding of these markers to enhance prenatal care and facilitate targeted interventions

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria specified pregnant women aged 20 to 40, diagnosed with preeclampsia based on blood pressure and proteinuria

Exclusion Criteria:

* applied to those with diabetes, liver or kidney diseases, cardiovascular diseases, or using specific supplements like vitamins A, C, and E.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study population, comprising preeclamptic and healthy pregnant women, was meticulously defined using anthropometric questionnaires and consideration of relevant medical features
Study Population: 45 with preeclampsia who completed the questionnaire, providing all necessary data
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Oxadative stress parameters | 7 months
  Thioredoxin and 4-Hydroxynonenal quantification, while malondialdehyde
Thioredoxin and 4-Hydroxynonenal quantification, while malondialdehyde | 7 months
  Thioredoxin and 4-Hydroxynonenal quantification, while malondialdehyde

OTHER OUTCOMES:
Preeclampsia parameters | 7 months
  Total cholesterol (TC), random blood glucose (RBG), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)

CONTACTS AND LOCATIONS:
Overall Officials: Doaa El-Bohy, PhD, Principal Investigator — Al-Ahliyya Amman University
Locations (1):
- Al-Ahliyya Amman University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Consent forms